CLINICAL TRIAL: NCT07131982
Title: The Effect of Watching Animation-Assisted Preoperative Informative Video Using Virtual Reality on Perioperative Anxiety and Fear in Children and Mothers: A Randomized Controlled Study
Brief Title: The Effect of Informative Animated Videos Watched Before Surgery on Anxiety and Fear in Children and Their Mothers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Yağmur Sezer Efe, Associate Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ERU-SBF-YZE-01
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Surgery in Children
Keywords: children; anxiety; surgery; fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: intervention group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): On the morning of the surgery, before the operation, children and their mothers who are included in the training group will be administered the following questionnaires: the Physiological Parameters Measurement Form, the Children's Fear Scale, and the Multidimensional Perioperative Anxiety Scale for Children (for children) and the State Anxiety Inventory-Short Form (for mothers). After the scales are administered, a pre-recorded video content, approximately 5 minutes in length and written by the researchers, will be shown to the child and mother on the morning of the surgery using a Virtual Reality Headset. Fifteen minutes after the video presentation, the Physiological Parameters Measurement Form, Multidimensional Perioperative Anxiety Scale for Children, and Children's Fear Scale will be administered to the children, and the State Anxiety Inventory-Short Form will be administered to the mothers. One hour post-op, the Physiological Parameters Measurement Form, Multidimensional Periop
  Interventions: Other: Informative Animated Video to be Viewed with Virtual Reality Glasses
- control group (No Intervention): No interventions other than clinical routines will be performed on children in the control group, and they will be evaluated during the standard care process. Before surgery, the Physiological Parameters Measurement Form, Children's Fear Scale, and Multidimensional Perioperative Anxiety Scale questions will be administered to children, and the State Anxiety Inventory-Short Form questions will be administered to mothers. The scales will be administered again 15 minutes after administration and at the 1-hour post-operative mark.

INTERVENTIONS:
Other: Informative Animated Video to be Viewed with Virtual Reality Glasses — No study has been found in the literature evaluating the effect of animated videos shown to children through virtual reality glasses on mothers and children. The aim of this study was to determine the effect of animated videos shown through virtual reality glasses before surgery on perioperative anxiety and fear in children and their mothers.
  Arms: intervention group

SUMMARY:
It is important to prepare children and their mothers psychologically for surgery. There are many initiatives to achieve this psychological preparation, including interactive educational booklets for children and their families, hospital tours, educational multimedia applications, web-based preparation programs, virtual reality applications, virtual tours, therapeutic games, hospital clowning, and educational coloring books. Among these initiatives, the immersive features of virtual reality glasses are seen as an effective method for distracting children from negative stimuli. Informing children before surgery is effective in increasing their sense of control during medical and surgical interventions. The information provided before surgery effectively reduces pain and fear in children. This research aims to reduce the anxiety and fear of children undergoing surgery and their mothers, as well as to facilitate the child's recovery after surgery. Additionally, reducing the mother's anxiety and fear will enable her to provide higher-quality care to her child during the postoperative process.

This study will be conducted using a prospective randomized controlled study design, matching children according to gender, age, and minor surgical reason, to determine the effect of animated videos shown through virtual reality glasses before surgery on perioperative anxiety and fear in children and their mothers.

The objectives of the study are:

* The animated video to be shown will reduce children's and mothers' fear of surgery.
* The animated video to be shown will reduce children's and mothers' perioperative anxiety.

DETAILED DESCRIPTION:
Surgical procedures are difficult experiences that create stress and anxiety for children and their families. Children's dependence on others to fulfill their roles during the hospital stay and surgery can lead to a loss of control and anxiety. Furthermore, the disruption of physical integrity, pain, and discomfort can lead to stress and anxiety in children and their parents. Parental stress often manifests as anxiety, anger, fear, or apprehension. Children affected by their mothers' anxiety, who are their primary caregivers, may fear something bad will happen to them or that something is being hidden from them. Children's anxiety about surgery can lead to postoperative behavioral problems such as separation anxiety, eating disorders, nightmares, and enuresis.

Reducing children's anxiety in the preoperative period is crucial to preventing negative postoperative outcomes. Preparations for this include interactive educational booklets, hospital tours, educational multimedia applications, web-based preparation programs, virtual reality applications, virtual tours, therapeutic games, hospital clowning, and educational coloring books, among many other initiatives. Among these interventions, the immersive features of virtual reality headset technology are seen as an effective method for distracting children from negative stimuli. Virtual reality slows down the response to pain and anxiety in children. Recent studies have used virtual reality headsets to increase children's comfort and familiarity with medical procedures and treatment environments, and technology-based preoperative preparation interventions have been reported to be effective in alleviating preoperative anxiety in children. The literature contains research findings on the effectiveness or ineffectiveness of methods used to reduce preoperative anxiety and fear in children. However, no studies have been found that evaluate the effects of animated videos shown to children on mothers and children. The purpose of this study was to determine the effect of animated videos viewed through virtual reality headsets before surgery on perioperative anxiety and fear in children and their mothers.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-13,
* Those who will undergo surgery for the first time,
* Able to read and write,
* Her mother and herself agreed to participate in the study,
* No communication problems,
* It will be done with children who can speak and understand Turkish and their mothers.

Exclusion Criteria:

* With developmental disabilities,
* Having a history of neurological disease or psychoactive drug use,
* Those with hearing and/or visual impairments,
* Children with a history of previous surgery and their mothers will not be included in the study.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-12-11 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Perioperative Anxiety Scale for Children | one month
  This scale was developed by Chow and colleagues to assess perioperative anxiety in children aged 7-13 years undergoing day surgery. As the score increases, anxiety increases. The scale is administered to children aged 7-13 years a total of three times: on the day the surgical procedure date is scheduled, on the day of the surgical procedure, and one month after the surgical procedure.

SECONDARY OUTCOMES:
Child Fear Scale | one month
  The Children's Fear Scale, developed by McMurtry and colleagues, is used to measure children's fears and anxieties.As the score increases, fear increases
State-trait Anxiety Inventory | one month
  A form that measures state anxiety and trait anxiety. As the score increases, state-trait anxiety increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No